CLINICAL TRIAL: NCT03473951
Title: The Dose-response Effect of Serum Uric Acid on the Prevalence and Electrocardiographic Left Ventricular Hypertrophy in the Apparently Healthy Individuals
Brief Title: The Relationship Among, Serum Uric Acid, Left Ventricular Hypertrophy and Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Cheng-Wei Liu, Cardiologist, National Defense Medical Center, Taiwan
Other Study IDs: 2-106-05-148
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Hyperuricemia; Healthy
Keywords: Hyperuricemia; Metabolic syndrome; Left ventricular hypertrophy
MeSH Terms: conditions — Hyperuricemia; Metabolic Syndrome; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperuricemia: Hyperuricemia is defined as a serum uric acid level of 7 mg/dl or more in men or 6 mg/dl or more in women
  Interventions: Diagnostic Test: Hyperuricemia

INTERVENTIONS:
Diagnostic Test: Hyperuricemia — Hyperuricemia vs. normouricemia

SUMMARY:
Hyperuricemia is associated with the prevalence of metabolic syndrome and cardiovascular risks in diverse of the population. Whether the dose-response effects on the prevalence of metabolic syndrome and cardiometabolic risks is unclear. The present study is conducted to investigate the relationship between serum uric acid and the prevalence metabolic syndrome and left ventricular hypertrophy.

DETAILED DESCRIPTION:
Apparently healthy individuals with an estimated screening number of approximately twenty-thousand individuals undergo an annual health exam in the investigators' hospital. The routine exam includes measurements of body height, body weight, blood pressure, visual and acoustic acuity, physical examinations, basic blood tests, urine analyses, chest radiography, and electrocardiography. The blood tests were performed after individuals fasted for at least eight hours. Individuals with any abnormal results underwent a clinical examination at an outpatient department for safety issues, ensuring the accuracy of the data. All data were registered prospectively. The investigators retrospectively collected data from the annual exam.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ages of 20-65 years underwent the annual health exam at the investigators' hospital.

Exclusion Criteria:

* The individual had no data to define metabolic syndrome, including waist circumference, office blood pressure, serum uric acid, triglyceride, high-density lipoprotein cholesterol, fasting glucose.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy individuals routinely underwent the annual health exam.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of metabolic syndrome | 1 day
  Based on the Taiwan criteria, metabolic syndrome must fulfill at least three of the five following criteria: 1) waist circumference more than 90 cm in men or more than 80 cm in women; 2) blood pressure of more than 130 / 85 mm Hg or already on anti-hypertensive medication; 3) fasting glucose of 100 mg/dl or more or already on anti-diabetic agents; 4) triglyceride level of 150 mg/dl or more or already on lipid lowering therapy for hypertriglyceridemia; 5) high-density lipoprotein cholesterol of 40 mg/dl or less in men or 50 mg/dl or less in women; the investigators also replaced the criterion of waist circumference by body mass index of 27 kg/m2 in the definition of metabolic syndrome.

SECONDARY OUTCOMES:
Left ventricular hypertrophy - Cornell voltage criteria. | 1 day
  Left ventricular hypertrophy is defined by Cornell voltage criteria.
Left ventricular hypertrophy - Cornell voltage product. | 1 day
  Left ventricular hypertrophy is defined by Cornell voltage product.
Left ventricular hypertrophy - Sokolow-Lyon criteria. | 1 day
  Left ventricular hypertrophy is defined by Sokolow-Lyon criteria.
Left ventricular hypertrophy - Minnesota Code electrocardiographic classification. | 1 day
  Left ventricular hypertrophy is defined by Minnesota Code electrocardiographic classification.
Left ventricular hypertrophy - composite of Cornell voltage criteria, Cornell voltage product, Sokolow-Lyon criteria, Minnesota Code electrocardiographic classification. | 1 day
  Any of above left ventricular hypertrophy criteria is counted as left ventricular hypertrophy.
brief symptom rating scale-5 | 1 day
  Brief symptom rating scale-5 consisted of five items with a total score of 0 to 20. Each items range from 0 to 4 in score, including difficult in falling asleep, anxiety (feeling tense or high-strung), hostility (feeling easily annoyed or irritated), interpersonal sensitivity (feeling inferior to others), depression (feeling depressed or in a low mood) in the past week. The summation of brief symptom rating scale-5 is further classified as normal (score of <6), mild mood disorder (score of 6-9), moderate mood disorder (score of 10-14), severe mood disorder (score of >14). Suicidal attempt is an additional item and the score >1 is considered as severe mood disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service General Hospital, songshan branch, Taipei, Songshan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tu CM, Wei TE, Tseng GS, Chen CC, Liu CW. Serum uric acid is associated with incident metabolic syndrome independent of body shape index and body roundness index in healthy individuals. Nutr Metab Cardiovasc Dis. 2021 Oct 28;31(11):3142-3151. doi: 10.1016/j.numecd.2021.07.008. Epub 2021 Jul 24. PMID 34518090
- [Derived] Liu CW, Ke SR, Tseng GS, Wu YW, Hwang JJ. Elevated serum uric acid is associated with incident hypertension in the health according to various contemporary blood pressure guidelines. Nutr Metab Cardiovasc Dis. 2021 Apr 9;31(4):1209-1218. doi: 10.1016/j.numecd.2021.01.003. Epub 2021 Jan 12. PMID 33618920
- [Derived] Liu CW, Chen KH, Tseng CK, Chang WC, Wu YW, Hwang JJ. The dose-response effects of uric acid on the prevalence of metabolic syndrome and electrocardiographic left ventricular hypertrophy in healthy individuals. Nutr Metab Cardiovasc Dis. 2019 Jan;29(1):30-38. doi: 10.1016/j.numecd.2018.10.001. Epub 2018 Oct 16. PMID 30545672